CLINICAL TRIAL: NCT06850883
Title: A Simulation Training Program for Person-Centered In-Home Dementia Care
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: National Taipei University of Nursing and Health Sciences (Other)
Responsible Party: Principal Investigator, Li-Min Kuo, Associate Professor, National Taipei University of Nursing and Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NSTC 113-2314-B-227-005 -
Record Dates: First submitted 2025-02-19; First posted 2025-02-27 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Dementia
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A person-centered dementia home care scenario-based training program (Experimental)
  Interventions: Other: A person-centered dementia home care scenario-based training program
- control arm (Placebo Comparator)
  Interventions: Other: Routine Treatment

INTERVENTIONS:
Other: A person-centered dementia home care scenario-based training program — The training program primarily consists of three major themes in dementia care scenario-based training: "Empathy," "Challenging Behavior Management," and "Interactive Activity Design."
  Arms: A person-centered dementia home care scenario-based training program
Other: Routine Treatment — Routine Treatment
  Arms: control arm

SUMMARY:
This study primarily explores the impact of a person-centered dementia home care scenario-based training program on home care workers' empathy, care preparedness, competence, predictability, and rewards.

ELIGIBILITY:
Inclusion Criteria:

(A) Aged 20 years or older; (B) Employed as a full-time worker in a home-based long-term care service institution; (C) Willing to participate in this study.

Exclusion Criteria:

* Employed as a part-time worker in a home-based long-term care service institution

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-03-15 (Actual); Primary Completion 2025-03-15 (Actual); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
Empathy Level in Formal Caregivers | pretest, Immediately after intervention, 1 month after intervention completion
  Measured using the Jefferson Scale of Empathy, with scores ranging from 20 to 140. Higher scores indicate greater empathy.
Preparedness Level in Formal Caregivers | pretest, Immediately after intervention, 1 month after intervention completion
  Measured using the Archbold Scale of Preparedness, with mean scores ranging from 0 to 4. Higher scores indicate greater Preparedness.
Competence Level in Formal Caregivers | pretest, Immediately after intervention, 1 month after intervention completion
  Measured using the Kosbery and Caril Scale of Competence, with mean scores ranging from 1 to 5. Higher scores indicate greater Competence.
Predictability Level in Formal Caregivers | pretest, Immediately after intervention, 1 month after intervention completion
  Measured using the Levine Scale of Predictability, with mean scores ranging from 0 to 4. Higher scores indicate greater Predictability.
Rewards Level in Formal Caregivers | pretest, Immediately after intervention, 1 month after intervention completion
  Measured using the Archbold Scale of Rewards, with mean scores ranging from 0 to 4. Higher scores indicate greater Rewards.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taipei University of Nursing and Health Sciences, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No